CLINICAL TRIAL: NCT00760513
Title: The Effects of Purified n-3 Fatty Acids on Serum Fibrosis Markers and Cardiovascular Risk Markers in a Randomized Placebo Controlled Trial in Patients With Non Alcoholic Fatty Liver Disease
Brief Title: Treatment of Non Alcoholic Fatty Liver Disease With n-3 Fatty Acids
Acronym: WELCOME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-12-59. (R&D: RHM MED 0836); 08/H0502/165 (Other: Local Research Ethics Committee)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: non alcoholic fatty liver disease; NAFLD; fish oil; intervention; RCT; biomarkers
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Omacor

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega 3 fatty acid (fish oil) (Active Comparator): OMACOR (alternative name: Lovaza) 4 grammes daily, oral capsule
  Interventions: Drug: OMACOR
- dummy pill (Placebo Comparator): 4 grammes daily, oral capsule (olive oil)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: OMACOR — 4 grammes daily, oral capsule
  Other Names: Lovaza
  Arms: Omega 3 fatty acid (fish oil)
Drug: Placebo oral capsule — 4 grammes daily, oral capsule (olive oil)
  Other Names: Dummy
  Arms: dummy pill

SUMMARY:
Non alcoholic fatty liver disease (NAFLD) imposes a high and increasing burden on the NHS, yet there is presently no licensed treatment or validated approach to management. NAFLD predisposes to increased risk of type 2 diabetes, increased risk of cardiovascular disease and may progress to chronic irreversible liver disease.

In NAFLD patients, the investigators will test the hypothesis that treatment with long chain n-3 fatty acid supplementation for 18 months favourably influences bio-markers for NAFLD and risk factors for cardiovascular disease and type 2 diabetes.

DETAILED DESCRIPTION:
We will recruit people with NAFLD who have been diagnosed as part of their NHS care with having this condition. At present there is no treatment for this condition. Over time a proportion of people with NAFLD.

Purpose and design

We are asking the research question ' Does treatment with purified long chain n-3 fatty acids (purified fish oil) improve non alcoholic fatty liver disease and risk factors for heart disease and type 2 (adult) diabetes that are strongly linked to this liver condition?'

Presently there is no treatment for this liver condition. Research evidence suggests that purified long chain n-3 fatty acids might be beneficial for this condition.

To address this research question we want to undertake a randomised double blind placebo controlled trial recruiting people who have been diagnosed with a liver biopsy as having the liver condition.

A protocol change that were approved during in the course of the study in October 2011.

In the protocol, we have deleted information regarding liver biopsy that was to be offered at the end of the study.

Having collated volunteer opinion and local consultant opinion, whereas a high proportion of volunteers were happy to undergo a follow up liver biopsy, our local hepatologists now consider that in 2011, the small risk of morbidity and mortality of volunteers undergoing liver biopsy is unacceptable, within the context of a research study. Their opinions have changed since 2008 when the initial LREC approval was granted.

Liver biopsy was always an optional extra and would only have been undertaken in a subgroup of the volunteers. Therefore, removal of liver biopsy from the protocol does not affect the validity of the study to test effects of the n-3 fatty acid intervention on biomarkers and liver fat in people with non alcoholic fatty liver disease.

Besides removal of liver biopsy from the protocol, we have clarified in the protocol, the end points of the study and numbers randomised to either n-3 fatty acid or placebo (n=100, as always intended). We have also made it clear in the amendment that measurement of liver fat is also a primary outcome of the study. (We already have permission to undertake this test but it was uncertain when the study was approved that we would have sufficient funding for this expensive test and it was originally not a primary outcome).

We have therefore added a power calculation (and cited the relevant literature) to show that with a sample size of n=100 people, based upon the known treatment effects of n-3 fatty acids on liver fat, we have acceptable power to detect the predicted decrease in this outcome with treatment.

ELIGIBILITY:
Inclusion criteria:

1. Steatohepatitis diagnosed on normal clinical grounds including in most cases liver biopsy and assessed by Kleiner scoring system to assess severity, with no known aetiological factors for underlying liver disease (e.g. exclusion of hepatitis A, B & C, primary biliary cirrhosis, autoimmune hepatitis, haemochromatosis).
2. Steatosis diagnosed by ultrasound, CT or magnetic resonance imaging who also have either diabetes and/or features of the metabolic syndrome, without evidence of known aetiological factors for underlying liver disease (e.g. exclusion of hepatitis A, B & C, primary biliary cirrhosis, autoimmune hepatitis, haemochromatosis).

Liver biopsy or liver scan will be within 3 years of recruitment to the study. Age: men & women >18 years. Alcohol consumption <35 units / week for women <50 units / week for men).

Exclusion criteria:

* Decompensated acute or chronic liver disease, or harmful drinking (> 35 u/week in women > 50 u /week in men).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2013-11-01 (Actual); Study Completion 2018-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Byrne, MBBCh PhD, Principal Investigator — University of Southampton, UK
Locations (1):
- Southamption General Hospital, Southampton, Hants, United Kingdom

REFERENCES:
- [Background] Scorletti E, Bhatia L, McCormick KG, Clough GF, Nash K, Calder PC, Byrne CD; WELCOME Trial Investigators. Design and rationale of the WELCOME trial: A randomised, placebo controlled study to test the efficacy of purified long chainomega-3 fatty acid treatment in non-alcoholic fatty liver disease [corrected]. Contemp Clin Trials. 2014 Mar;37(2):301-11. doi: 10.1016/j.cct.2014.02.002. Epub 2014 Feb 18. PMID 24556343
- [Background] Guha IN, Parkes J, Roderick P, Chattopadhyay D, Cross R, Harris S, Kaye P, Burt AD, Ryder SD, Aithal GP, Day CP, Rosenberg WM. Noninvasive markers of fibrosis in nonalcoholic fatty liver disease: Validating the European Liver Fibrosis Panel and exploring simple markers. Hepatology. 2008 Feb;47(2):455-60. doi: 10.1002/hep.21984. PMID 18038452
- [Background] Angulo P, Hui JM, Marchesini G, Bugianesi E, George J, Farrell GC, Enders F, Saksena S, Burt AD, Bida JP, Lindor K, Sanderson SO, Lenzi M, Adams LA, Kench J, Therneau TM, Day CP. The NAFLD fibrosis score: a noninvasive system that identifies liver fibrosis in patients with NAFLD. Hepatology. 2007 Apr;45(4):846-54. doi: 10.1002/hep.21496. PMID 17393509
- [Result] Scorletti E, Bhatia L, McCormick KG, Clough GF, Nash K, Hodson L, Moyses HE, Calder PC, Byrne CD; WELCOME Study. Effects of purified eicosapentaenoic and docosahexaenoic acids in nonalcoholic fatty liver disease: results from the Welcome* study. Hepatology. 2014 Oct;60(4):1211-21. doi: 10.1002/hep.27289. PMID 25043514
- [Derived] Hodson L, Bhatia L, Scorletti E, Smith DE, Jackson NC, Shojaee-Moradie F, Umpleby M, Calder PC, Byrne CD. Docosahexaenoic acid enrichment in NAFLD is associated with improvements in hepatic metabolism and hepatic insulin sensitivity: a pilot study. Eur J Clin Nutr. 2017 Aug;71(8):973-979. doi: 10.1038/ejcn.2017.9. Epub 2017 Mar 15. PMID 28294174
- [Derived] Clough GF, McCormick KG, Scorletti E, Bhatia L, Calder PC, Griffin MJ, Byrne CD. Higher body fat percentage is associated with enhanced temperature perception in NAFLD: results from the randomised Wessex Evaluation of fatty Liver and Cardiovascular markers in NAFLD with OMacor thErapy trial (WELCOME) trial. Diabetologia. 2016 Jul;59(7):1422-1429. doi: 10.1007/s00125-016-3966-8. Epub 2016 Apr 22. PMID 27106721
- [Derived] Bhatia L, Scorletti E, Curzen N, Clough GF, Calder PC, Byrne CD. Improvement in non-alcoholic fatty liver disease severity is associated with a reduction in carotid intima-media thickness progression. Atherosclerosis. 2016 Mar;246:13-20. doi: 10.1016/j.atherosclerosis.2015.12.028. Epub 2015 Dec 24. PMID 26748347
- [Derived] Byrne CD, Targher G. Time to Replace Assessment of Liver Histology With MR-Based Imaging Tests to Assess Efficacy of Interventions for Nonalcoholic Fatty Liver Disease. Gastroenterology. 2016 Jan;150(1):7-10. doi: 10.1053/j.gastro.2015.11.016. Epub 2015 Nov 18. No abstract available. PMID 26602219
- [Derived] Scorletti E, West AL, Bhatia L, Hoile SP, McCormick KG, Burdge GC, Lillycrop KA, Clough GF, Calder PC, Byrne CD. Treating liver fat and serum triglyceride levels in NAFLD, effects of PNPLA3 and TM6SF2 genotypes: Results from the WELCOME trial. J Hepatol. 2015 Dec;63(6):1476-83. doi: 10.1016/j.jhep.2015.07.036. Epub 2015 Aug 10. PMID 26272871
- [Derived] McCormick KG, Scorletti E, Bhatia L, Calder PC, Griffin MJ, Clough GF, Byrne CD. Impact of high dose n-3 polyunsaturated fatty acid treatment on measures of microvascular function and vibration perception in non-alcoholic fatty liver disease: results from the randomised WELCOME trial. Diabetologia. 2015 Aug;58(8):1916-25. doi: 10.1007/s00125-015-3628-2. Epub 2015 May 29. PMID 26021488
- [Derived] Byrne CD, Targher G. Ectopic fat, insulin resistance, and nonalcoholic fatty liver disease: implications for cardiovascular disease. Arterioscler Thromb Vasc Biol. 2014 Jun;34(6):1155-61. doi: 10.1161/ATVBAHA.114.303034. Epub 2014 Apr 17. PMID 24743428
- [Derived] Targher G, Byrne CD. Clinical Review: Nonalcoholic fatty liver disease: a novel cardiometabolic risk factor for type 2 diabetes and its complications. J Clin Endocrinol Metab. 2013 Feb;98(2):483-95. doi: 10.1210/jc.2012-3093. Epub 2013 Jan 4. PMID 23293330

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omega 3 Fatty Acid (Fish Oil) | Dummy Pill
Started | 51 | 52
Completed | 46 | 45
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega 3 Fatty Acid (Fish Oil) | Dummy Pill | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 46 | 93
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (11.1) | 54 (9.6) | 51.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 17 | 43
  Male | 25 | 35 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 51 | 52 | 103

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Liver Fat
Description: Percentage of liver fat was measured using magnetic resonance spectroscopy at baseline and end of study. High percentage values indicate a lot of liver fat (scale from 0 to 100%). Change in liver fat percentage represented the arithmetical difference between end of study liver fat percentage minus baseline measurement of liver fat percentage change in liver fat percentage was used to test whether the intervention decreased liver fat percentage. A negative change value in liver fat percentage indicates a response to therapy. A positive change value indicates no response to therapy.
Time Frame: Baseline and 18 months
Measure: Mean (Standard Deviation); unit: percentage of liver fat
Arm/Group | Omega 3 Fatty Acid (Fish Oil) | Dummy Pill
Number analyzed (Participants) | 46 | 45
percentage of liver fat | -7.9 (17.4) | -4.6 (9.2)
Statistical Analysis 1: Comparison: Omega 3 Fatty Acid (Fish Oil) vs Dummy Pill; We estimated that a 20% decrease in liver fat with Omacor treatment, assuming a sigma of 0.3, and an alpha of 0.05; with 91 participants completing our trial, we had 86% power to detect a 20% change in liver fat (two tailed test) (see HEPATOLOGY 2014;60:1211-1221); Test type: Superiority; p = 0.48, Regression, Linear — The a priori threshold for statistical significance = P</=0.05; Adjusted for baseline value of liver fat percentage; Mean Difference (Net) = -1.7, 95% CI 2-sided [-6.3 to 3.0]

2. Primary Outcome: Liver Fibrosis Score
Description: The Liver Fibrosis Score is an algorithmically derived score of liver fibrosis comprising measurements of tissue matrix metalloproteinase-1 (TIMP-1), hyaluronic acid (HA) and the amino terminal end of procollagen III (PIIINP) (see Guha et al. in Reference section). The Score represents a number on a numerical scale from 0 to 20. High values of the score (measured in arbitrary units) indicate high probability of advanced liver fibrosis, low scores indicate low probability of advanced liver fibrosis. Change in Liver Fibrosis Score was used to test the intervention. Change in liver fibrosis score represented the change in measurement as calculated as the arithmetic difference between the end value minus the baseline value of the Liver Fibrosis Score. The change in Liver Fibrosis Score can therefore be negative (representing an improvement in liver fibrosis between baseline and end of study) or be positive, (representing a worsening a liver fibrosis between baseline and end of study.
Time Frame: Baseline and 18 months
Population: Participants with baseline and end of study data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega 3 Fatty Acid (Fish Oil) | Dummy Pill
Number analyzed (Participants) | 46 | 45
score on a scale | 0.3 (0.6) | 0.2 (0.6)
Statistical Analysis 1: Comparison: Omega 3 Fatty Acid (Fish Oil) vs Dummy Pill; Based on the available evidence at the time, we assumed that a 0.6-1.0 unit change in fibrosis score might be clinically significant (Hepatology 2008 Feb;47(2):455-460). Consequently, to detect a minimum 0.6 unit change in score (e.g. 9.0 at baseline and 8.4 at the end of the study) with an SD of 1.0, 100 participants would provide >80% power at the 5% significance level, and with a 15% drop out of participants there would also be >80% power to detect this effect; Test type: Superiority; p = 1.0, Regression, Linear — A priori p value threshold </=0.5; Adjusted for baseline; Mean Difference (Net) = -0.001, 95% CI 2-sided [-0.3 to 0.3]

3. Primary Outcome: NAFLD Fibrosis Score
Description: The NAFLD fibrosis score represented a validated algorithmically-derived measure of liver fibrosis as reported in Angulo et al (see reference section). The Score is derived from anthropometric and biochemical measurements in subjects. The NAFLD fibrosis score represents an arbitrary number with no units from -5.0 to +5.0. High positive NAFLD fibrosis scores indicate a high probability of advanced liver fibrosis. Negative scores represent a low probability of advanced liver fibrosis. The change in NAFLD fibrosis score (measured in arbitrary units) was used to test the effect of the intervention and represented the arithmetic difference in the end minus baseline measurements of this score. Thus, a negative change in the Score in the Table represented an improvement in liver fibrosis score between baseline and the end of the study. A positive change in the Score in the Table represented a worsening in liver fibrosis score between baseline and end of the study.
Time Frame: Baseline and 18 months
Population: Participants with baseline and end of study data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega 3 Fatty Acid (Fish Oil) | Dummy Pill
Number analyzed (Participants) | 46 | 45
score on a scale | 0.8 (0.9) | 0.8 (0.7)
Statistical Analysis 1: Comparison: Omega 3 Fatty Acid (Fish Oil) vs Dummy Pill; There was no power calculation for this end point; Test type: Superiority; p = 0.9, Regression, Linear — A priori threshold for statistical significance p </=0.05; Adjusted for baseline measurement; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.4 to 0.3]

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- Dummy Pill: 4 grammes daily, oral capsule (olive oil)
  OMACOR: 4 grammes daily, oral capsule
Arm/Group | Omega 3 Fatty Acid (Fish Oil) | Dummy Pill
Serious Adverse Events (participants affected / at risk) | 4/51 | 8/52
Other Adverse Events (participants affected / at risk) | 49/51 | 44/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omega 3 Fatty Acid (Fish Oil) (N=51) | Dummy Pill (N=52)
Anaemia and disorientation (Gastrointestinal disorders) | 1 | 0
seminoma (Surgical and medical procedures) | 0 | 1
cellulitis on right lateral malleolus (Skin and subcutaneous tissue disorders) | 1 | 0
Acute asthma attack (Respiratory, thoracic and mediastinal disorders) | 0 | 1
stabilisation of her diabetes (Endocrine disorders) | 0 | 1
severe chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laparoscopy and appendectomy (Surgical and medical procedures) | 0 | 1
chest pain radiating to the neck with tingling to left arm (Cardiac disorders) | 0 | 1
laparoscopic adhesiolysis (Surgical and medical procedures) | 0 | 1
elective hysterectomy (Surgical and medical procedures) | 0 | 1
removal of myxoma (Surgical and medical procedures) | 0 | 1
Tonsillectomy (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omega 3 Fatty Acid (Fish Oil) (N=51) | Dummy Pill (N=52)
dermatological disorders (Skin and subcutaneous tissue disorders) | 8 | 9
Nausea and vomitting (Gastrointestinal disorders) | 3 | 4
accidental fall (General disorders) | 0 | 2
achile's heel and foot problems (General disorders) | 0 | 2
anaemia (Blood and lymphatic system disorders) | 2 | 0
anxiety and depression (General disorders) | 4 | 2
asthma and breathing (Respiratory, thoracic and mediastinal disorders) | 3 | 0
back pain and sciatica (Musculoskeletal and connective tissue disorders) | 3 | 2
carpal disorders (Musculoskeletal and connective tissue disorders) | 0 | 1
urological disorders (Renal and urinary disorders) | 5 | 11
chest infection (Infections and infestations) | 13 | 4
chest pain and ecg alterations (Cardiac disorders) | 5 | 5
dental disorders (General disorders) | 0 | 2
diarrhea (Gastrointestinal disorders) | 4 | 6
dyslipidaemia (Metabolism and nutrition disorders) | 1 | 1
fall and fracture (General disorders) | 1 | 0
fertility problems (Reproductive system and breast disorders) | 1 | 0
fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
flu, cough and sore throat (Respiratory, thoracic and mediastinal disorders) | 13 | 5
fluid retention and oedema (General disorders) | 0 | 2
gastrointestinal disorder (Gastrointestinal disorders) | 6 | 5
gynecological disorders (Reproductive system and breast disorders) | 2 | 1
headache and dizziness (General disorders) | 6 | 6
hepatological disorder (Hepatobiliary disorders) | 0 | 1
hyperglycaemia & hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3
hypertension (General disorders) | 5 | 1
insomnia (General disorders) | 1 | 0
joint pain (Musculoskeletal and connective tissue disorders) | 13 | 11
knee surgery (Musculoskeletal and connective tissue disorders) | 2 | 0
liver biopsy (Hepatobiliary disorders) | 1 | 0
neurological disorders (Nervous system disorders) | 1 | 0
onset diabetes (Endocrine disorders) | 2 | 1
ophtalmological disorders (Eye disorders) | 0 | 6
orthopedic disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
other drug overdose (Product Issues) | 2 | 0
other drug reaction (Product Issues) | 5 | 0
otolaryngological disorders (Ear and labyrinth disorders) | 10 | 3
pregnancy (Reproductive system and breast disorders) | 1 | 0
proctological disorders (Gastrointestinal disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes